CLINICAL TRIAL: NCT05974189
Title: Assessing Vericiguat for the Management of Heart Failure With Reduced Ejection Fraction Using HealthVerity Data
Brief Title: The VERIFY Study: An Observational Study Called VERIFY to Learn More About the Use of Vericiguat in People With Chronic Heart Failure With Reduced Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22562
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFrEF patients treated with at least one GDMT and with vericiguat: This study will use anonymized real-world data from HealthVerity closed Medical and Pharmacy Claims.
  Adult patients with a diagnosis of HFrEF and received vericiguat added to at least one guideline directed medical therapy (GDMT), from January 1, 2021 through June 30, 2023 will be included in this retrospective cohort analysis.
- HFrEF patients treated with at least one GDMT, without vericiguat: This study will use anonymized real-world data from HealthVerity closed Medical and Pharmacy Claims.
  Adult patients with a diagnosis of HFrEF and received at least one GDMT (without vericiguat), from January 1, 2021 through June 30, 2023 will be included in this retrospective cohort analysis.

SUMMARY:
This is an observational study in which the health data of people with chronic heart failure with reduced ejection fraction (HFrEF) are collected using administrative claims data.

In observational studies, only observations are made and participants do not receive any advice or changes to healthcare.

Chronic HFrEF is a longterm condition that occurs when the heart is weak and cannot pump enough blood to the rest of the body with each heartbeat. This leads to a reduced supply of oxygen which the body requires to function properly. The common symptoms include breathlessness, weakness, fatigue, and swelling in the ankles and legs. If left untreated, heart failure can lead to other serious health problems, including damage to other organs, which may result in hospital stays and even death.

Vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC), which relaxes the blood vessels and allows more blood to flow through. As a result, the heart is able to pump better.

Vericiguat was approved for the treatment of HFrEF based on the results of a study called VICTORIA. The VICTORIA study showed that vericiguat helps in lowering the chances of death or hospitalization due to heart failure. There is limited information available about the use of vericiguat for the treatment of HFrEF under realworld conditions.

The main purpose of this study is to collect information about the characteristics of people with HFrEF, who are on vericiguat in addition to at least one standard treatment. Researchers will collect information about participants' basic characteristics, including their age, gender, other health conditions they may have, and the medicines they may be taking.

The data will come from administrative claims data for people in the United States of America who were diagnosed with HFrEF between January 2020 and June 2022.

In this study, only available data from routine care is collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-years old and have at least one year of continous enrollment in the HV database.
* Have proven or presumed HFrEF
* Have received ≥1 GDMTs for HFrEF
* All patients will be required to have continuous enrollment in the HealthVerity data set during the pre-index date (baseline period) of at least 90-days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort analysis in data from the deidentified, United States HealthVerity (HV) Claims, Pharmacy.
Sampling Method: Non-Probability Sample
Enrollment: 1391 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of baseline characteristics of new users administered vericiguat in addition to at least one GDMT in patients with HFrEF | Retrospective cohort analysis from 01-Jan-2018 to 30-Jun-2023

SECONDARY OUTCOMES:
First hospitalization for HF or all cause of death or first emergency room visit (ER) | Retrospective cohort analysis from 01-Jan-2018 to 30-Jun-2023
First ER visit or hospitalization for HF | Retrospective cohort analysis from 01-Jan-2018 to 30-Jun-2023
All-cause death | Retrospective cohort analysis from 01-Jan-2018 to 30-Jun-2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.